CLINICAL TRIAL: NCT01599325
Title: A Phase 2, Open-Label, Single-Arm Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Subcutaneous Azacitidine in Adult Chinese Subjects With Higher-Risk Myelodysplastic Syndromes
Brief Title: Study of Azacitidine to Evaluate Safety and Effectiveness for Chinese Patients With Higher Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA-MDS-002
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacitidine (Experimental): Azacitidine 75 mg/m^2/day subcutaneously (SC) for 7 days every 28 days until disease progression (DP), adverse events (AE), withdrawal of consent from further treatment, withdrawal of consent, death, lost to follow-up, or protocol violation.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Subcutaneous administration of azacitidine 75 mg/m^2/day for 7 days every 28 days optimally for at least 6 cycles until disease progression, unacceptable toxicity, or treatment discontinuation for any other reason
  Other Names: Vidaza

SUMMARY:
The purpose of the study is to determine whether azacitidine is safe and effective in the treatment of Chinese patients with higher risk Myelodysplastic Syndromes (MDS).

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

* Chinese males and females of Asian descent ≥ 18 years of age at the time of signing the informed consent document;
* Must have a documented diagnosis of refractory anemia with excess blasts (RAEB) or refractory anemia with excess blasts in transformation (RAEB-T) according to French-American-British (FAB) classification for Myelodysplastic Syndrome (MDS) and with an International Prognostic Scoring System (IPSS) score of intermediate-2 or high risk or a diagnosis of myelodysplastic chronic myelomonocytic leukemia (CMML) per modified FAB criteria meeting the following:

  * Monocytosis in peripheral blood > 1 x 10^9/L;
  * Dysplasia in one or more myeloid cell lines;
  * 10% to 29% blasts in the bone marrow; and White blood cell (WBC) count < 13 x 10^9/L
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 ;
* Adequate organ function, defined as:
* Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN);
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.0 times the ULN;
* Serum Creatinine ≤ 1.5 times the ULN;
* Females of childbearing potential (FCBP) must:
* Agree to the use of a physician-approved contraceptive method (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on azacitidine; and
* for 3 months following the last dose of azacitidine; and have a negative serum pregnancy test within 72 hours prior to starting Investigational Product (IP).
* Male subjects with a female partner of childbearing potential must agree to the use of a physician-approved contraceptive method throughout the course of the study and avoid fathering a child during the course of the study and for 3 months following the last dose of azacitidine;
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted;
* Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

* Previous treatment with azacitidine or decitabine;
* Diagnosis of malignant disease within the previous 12 months (excluding basal cell carcinoma of the skin without complications, "in-situ" carcinoma of the cervix or breast, or other local malignancy excised or irradiated with a high probability of cure);
* Uncorrected red cell folate deficiency or vitamin B12 deficiency;
* Diagnosis of metastatic disease;
* Malignant hepatic tumors;
* Known or suspected hypersensitivity to azacitidine or mannitol;
* Candidate to proceed to bone marrow or stem cell transplant during the study;
* Prior transplantation or cytotoxic therapy, including azacitidine and chemotherapy, administered to treat MDS;
* Treatment with erythropoietin or myeloid growth factors (granulocyte colony-stimulating factor [G-CSF] or granulocyte-macrophage colony-stimulating factor [GM-CSF]) during the 21 days prior to Day 1 of Cycle 1;
* Treatment with androgenic hormones during the 14 days prior to Day 1 of Cycle 1;
* Active viral infection with known human immunodeficiency virus (HIV) or viral hepatitis type B or C;
* Treatment with other investigational drugs, including thalidomide and arsenic trioxide, within the previous 30 days prior to Day 1 of Cycle 1, or ongoing adverse events from previous treatment with investigational drugs, regardless of the time period; and
* Pregnant or lactating females;
* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study;
* Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study;
* Any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-07-24 (Actual); Primary Completion 2015-01-29 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C L Beach, Study Director — Celgene
Locations (11):
- China (11):
  - Peking University People's Hospital, Beijing
  - The 301 Hospital- Chinese PLA General Hospital, Beijing
  - The Third Hospital of Peking University, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Guangdong General Hospital, Guangzhou
  - 1st Hospital Zhejiang University (The First Affiliated Hospital of Zhejiang University ), Hangzhou
  - Ruijin Hospital Shanghai Jiaotong University, Shanghai
  - Shanghai 6th Hospital, Shanghai
  - The 1st Hospital of Soochow University, Suzhou
  - Blood Disease Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Tianjin
  - Wuhan Union Hospital, Wuhan

RESULTS

PARTICIPANT FLOW:
Period: Primary Parent Phase
Arm/Group | Azacitidine
Started | 72
Intent to Treat (ITT) Population | 72 (Includes all participants who were enrolled into the study)
Pharmacokinetic (PK) Population | 12 (Includes all participants with evaluable azacitidine plasma PK profiles.)
Completed | 15 (Participants still on study treatment at time of study closure)
Not Completed | 57
Not completed — Adverse Event | 5
Not completed — Disease Progression | 7
Not completed — Withdrawal by Subject | 20
Not completed — Death | 13
Not completed — Protocol Violation | 1
Not completed — Lack of Therapeutic Effect | 9
Not completed — Other | 2
Period: Extension Phase
Arm/Group | Azacitidine
Started | 15
Completed | 0
Not Completed | 15
Not completed — Study Closure | 1
Not completed — Stopped to Receive Stem Cell Transplant | 1
Not completed — Lack of Therapeutic Effect | 4
Not completed — Disease Progression | 1
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Population: ITT includes all participants who had been screened and enrolled into the study.
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 38
International Prognostic Scoring System (IPSS) Risk Classification [Count of Participants; unit: Participants] — The Myelodysplastic Syndrome (MDS) IPSS score assesses the severity of MDS based on 3 prognostic factors each assigned a score: the percentage of bone marrow blasts, chromosome changes in the marrow cells (karyotype) and the presence of one or more low blood cell counts (cytopenias). The IPSS score is the sum of the bone marrow blast + karyotype + cytopenia score and ranges from 0 (low risk) to 3.5 (high risk). Prognosis is categorized as Low risk (score = 0), Intermediate-1 (score 0.5 to 1.0), Intermediate-2 (score 1.5 to 2.0) or High risk (score ≥ 2.5).
  Participants
    Low (0) | 0
    Intermediate 1 (0.5-1.0) | 0
    Intermediate 2 (1.5-2.0) | 47
    High (>=2.5) | 25
French-American-British classification (FAB) [Count of Participants; unit: Participants] — FAB is a classification system for five (5) subtypes of myelodysplastic syndrome that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts or a monocytosis. Classification was made by the Local Reviewer.
  Participants
    RAEB=Refractory anemia with excess blasts | 63
    RAEB in transformation | 8
    Modified CMML=Chronic myelomonocytic leukemia | 1
MDS World Health Organization (WHO) Classification [Count of Participants; unit: Participants] — The World Health Organization (WHO) classification recognizes eight subtypes of MDS that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts (i.e., erythroid precursors with iron deposits surrounding the nucleus), presence of a monocytosis or a deletion 5q.
  Participants
    RAEB-1=Refractory anemia with excess blasts | 14
    RAEB -2 with MPD=Myeloproliferative disease | 50
    Acute Myelogenous Leukemia (AML) | 7
    CMML | 1
    MDS and myeloproliferative disease (MPD) | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Hematologic Response Based on the International Working Group (IWG) Criteria for Myelodysplastic Syndrome (MDS) and Programmatically Assessed by the Sponsor Using Clinically Relevant Data.
Description: Hematologic Response is defined by those participants who experienced a Complete Response, Partial Response and Stable Disease (SD) based on IWG 2000 response criteria for MDS. CR = repeat bone marrow (BM) shows <5% myeloblasts, and peripheral blood values lasting ≥ 2 months of hemoglobin (hgb) (>110 g/L), neutrophils (≥1.5x10^9/L), platelets (≥100x10^9/L), blasts (0%) and no dysplasia • PR = same as CR for peripheral blood: BM shows blasts decrease by ≥ 50% or a less advanced FAB classification from pretreatment • Stable disease (SD): failure to achieve a PR, no evidence of progression for at least 2 months. • Failure: death during treatment or disease progression • Relapse After CR or PR: return to pretreatment BM blast percent or decrement of ≥ 50% from remission/response levels in granulocytes or platelets; or reduction in hgb by ≥20 g/L or transfusion dependence • Disease Progression: change in blast levels • Disease Transformation to Acute Myelogenous Leukemia.
Time Frame: Response initially assessed at end of cycle 6, then every 4 cycles; Up to 29 January 2015; 894 days
Population: Intent to Treat (ITT) includes all participants who were enrolled into the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
percentage of participants
  Overall CR+PR | 1.4 [0.0 to 7.5]
  Overall CR+PR+SD | 95.8 [88.3 to 99.1]
  Complete Remission (CR) | 1.4 [0.0 to 7.5]
  Partial Remission (PR) | 0 [0.0 to 5.0]

2. Primary Outcome: Percentage of Participants With a Hematologic Response Using IWG Criteria for MDS and Assessed by the Investigator
Description: as for outcome 1
Time Frame: Response initially assessed at end of cycle 6, then every 4 cycles; Up to 29 January 2015; 894 days
Population: Intent to Treat (ITT) includes all participants who were enrolled into the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
percentage of participants
  Overall CR+PR | 12.5 [5.9 to 22.4]
  Overall CR+PR+SD | 70.8 [58.9 to 81.0]
  CR | 6.9 [2.3 to 15.5]
  PR | 5.6 [1.5 to 13.6]

3. Primary Outcome: Percentage of Participants Achieving a Hematologic Improvement (HI) Based on 2000 IWG Response Criteria for MDS and Programmatically Assessed by the Sponsor Using Clinically Relevant Data.
Description: Hematologic improvements (HI) have 4 categories: 1. Erythroid response (HI-E): Major >20g/L increase or transfusion independent. Minor: 10-20g/L increase or ≥50% decrease in transfusion requirements. 2. Platelet response (HI-P): Major absolute increase of ≥30x10^9/L or platelet transfusion independence. Minor: ≥50% increase. 3. Neutrophil response (HI-N): Major 100% increase or an absolute increase of >0.5x10^9/L. Minor: ≥100% increase and absolute increase of <0.5x10^9/L 4. Progression or relapse after HI Hematological improvement (HI) was defined as any type (major or minor) of improvement of HI-E, HI-P, or HI-N. Criteria: Pretreatment=hemoglobin <100g/L or RBC transfusion-dependent, platelet count <100x10^9/L or platelet transfusion dependent, absolute neutrophil count <1.5x10^9/L. Sponsor's determination was derived using clinically relevant data. Denominator for progression/relapse after HI included participants who had achieved HI.
Time Frame: Up to 29 January 2015; 894 days
Population: Intent to Treat (ITT) includes all participants who were enrolled into the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
percentage of participants
  Any improvement | 52.8 [40.7 to 64.7]
  Hematologic Improvement-E (major) | 35.8 [24.5 to 48.5]
  Hematologic Improvement-E (minor) | 9.0 [3.4 to 18.5]
  Hematologic Improvement-P (major) | 37.9 [25.5 to 51.6]
  Hematologic Improvement-P (minor) | 0.0 [0.0 to 6.2]
  Hematologic Improvement-N (major) | 21.8 [11.8 to 35.0]
  Hematologic Improvement-N (minor) | 0.0 [0.0 to 6.5]

4. Secondary Outcome: The Number of Units of Platelet Transfusions by Cycle
Description: The number of units of platelet transfusions received 56 days prior to treatment, considered the baseline period, (baseline period defined as the screening period before the date of the first dose of azacitidine; any laboratory and blood transfusion data reported on the day of the first dose of azacitidine was considered to be baseline data) and during study was standardized per 28 days and summarized by cycle for platelets. The formula for standardizing per 28 days was: [(# of transfusions in the measurement period / length of the measurement period (days)) x 28], where the measurement period was either baseline or the relevant cycle length.
Time Frame: Up to cycle 27; The on-treatment period was considered the period from the date of first dose to the last treatment study visit; Up to 29 January 2015; 894 days
Population: Intent to Treat (ITT) includes all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: Units of platelet transfusions
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
Units of platelet transfusions
  Baseline N = 72 | 1.9 (4.91)
  Overall Post-Baseline Average N = 72 | 4.7 (17.79)
  Overall Change from Baseline N = 72 | 2.8 (17.89)
  Cycle 1 N = 72 | 5.2 (18.83)
  Cycle 2: number analyzed (Participants) | 66
  Cycle 2 | 2.4 (5.86)
  Cycle 3: number analyzed (Participants) | 59
  Cycle 3 | 3.3 (11.44)
  Cycle 4: number analyzed (Participants) | 56
  Cycle 4 | 2.7 (6.13)
  Cycle 5: number analyzed (Participants) | 50
  Cycle 5 | 2.5 (7.69)
  Cycle 6: number analyzed (Participants) | 46
  Cycle 6 | 1.5 (4.15)
  Cycle 7: number analyzed (Participants) | 39
  Cycle 7 | 1.0 (2.84)
  Cycle 8: number analyzed (Participants) | 36
  Cycle 8 | 1.1 (2.05)
  Cycle 9: number analyzed (Participants) | 31
  Cycle 9 | 0.8 (2.46)
  Cycle 10: number analyzed (Participants) | 29
  Cycle 10 | 0.8 (2.08)
  Cycle 11: number analyzed (Participants) | 28
  Cycle 11 | 0.5 (1.00)
  Cycle 12: number analyzed (Participants) | 24
  Cycle 12 | 0.3 (0.78)
  Cycle 13: number analyzed (Participants) | 17
  Cycle 13 | 0.3 (0.72)
  Cycle 14: number analyzed (Participants) | 15
  Cycle 14 | 0.1 (0.35)
  Cycle 15: number analyzed (Participants) | 13
  Cycle 15 | 0.3 (0.90)
  Cycle 16: number analyzed (Participants) | 10
  Cycle 16 | 0.3 (0.90)
  Cycle 17: number analyzed (Participants) | 7
  Cycle 17 | 0.3 (0.73)
  Cycle 18: number analyzed (Participants) | 7
  Cycle 18 | 0.6 (1.51)
  Cycle 19: number analyzed (Participants) | 6
  Cycle 19 | 0.3 (0.64)
  Cycle 20: number analyzed (Participants) | 4
  Cycle 20 | 0.2 (0.37)
  Cycle 21: number analyzed (Participants) | 3
  Cycle 21 | 0.0 (0.00)
  Cycle 22: number analyzed (Participants) | 1
  Cycle 22 | 0.0 (NA) — Not applicable = Null value
  Cycle 23: number analyzed (Participants) | 1
  Cycle 23 | 0.0 (NA) — Not applicable = Null value
  Cycle 24: number analyzed (Participants) | 1
  Cycle 24 | 0.0 (NA) — Not applicable = Null value
  Cycle 25: number analyzed (Participants) | 1
  Cycle 25 | 0.0 (NA) — Not applicable = Null value
  Cycle 26: number analyzed (Participants) | 1
  Cycle 26 | 0.0 (NA) — Not applicable = Null value
  Cycle 27: number analyzed (Participants) | 1
  Cycle 27 | 0.0 (NA) — Not applicable = Null value

5. Secondary Outcome: The Number of Platelet Transfusions by Cycle
Description: The number of platelet transfusions received 56 days prior to treatment, considered the baseline period (baseline period defined as the screening period before the date of the first dose of azacitidine; any laboratory and blood transfusion data reported on the day of the first dose of azacitidine was considered to be baseline data) and during study was standardized per 28 days and summarized by cycle for platelets. The formula for standardizing per 28 days was: [(# of transfusions in the measurement period / length of the measurement period (days)) x 28], where the measurement period was either baseline or the relevant cycle length.
Time Frame: as for outcome 4
Population: Intent to Treat (ITT) includes all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: Platelet transfusions
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
Platelet transfusions
  Baseline N = 72 | 0.8 (2.36)
  Overall Post-Baseline Average N = 72 | 1.6 (2.83)
  Overall Change from Baseline N = 72 | 0.8 (3.29)
  Cycle 1 N = 72 | 1.8 (2.89)
  Cycle 2: number analyzed (Participants) | 66
  Cycle 2 | 1.3 (2.59)
  Cycle 3: number analyzed (Participants) | 59
  Cycle 3 | 1.2 (2.28)
  Cycle 4: number analyzed (Participants) | 56
  Cycle 4 | 1.3 (2.18)
  Cycle 5: number analyzed (Participants) | 50
  Cycle 5 | 0.9 (1.58)
  Cycle 6: number analyzed (Participants) | 46
  Cycle 6 | 0.7 (1.34)
  Cycle 7: number analyzed (Participants) | 39
  Cycle 7 | 0.8 (2.50)
  Cycle 8: number analyzed (Participants) | 36
  Cycle 8 | 0.8 (1.66)
  Cycle 9: number analyzed (Participants) | 31
  Cycle 9 | 0.8 (2.46)
  Cycle 10: number analyzed (Participants) | 29
  Cycle 10 | 0.8 (2.08)
  Cycle 11: number analyzed (Participants) | 28
  Cycle 11 | 0.5 (1.00)
  Cycle 12: number analyzed (Participants) | 24
  Cycle 12 | 0.3 (0.78)
  Cycle 13: number analyzed (Participants) | 17
  Cycle 13 | 0.3 (0.72)
  Cycle 14: number analyzed (Participants) | 15
  Cycle 14 | 0.1 (0.35)
  Cycle 15: number analyzed (Participants) | 13
  Cycle 15 | 0.3 (0.90)
  Cycle 16: number analyzed (Participants) | 10
  Cycle 16 | 0.3 (0.90)
  Cycle 17: number analyzed (Participants) | 7
  Cycle 17 | 0.3 (0.73)
  Cycle 18: number analyzed (Participants) | 7
  Cycle 18 | 0.6 (1.51)
  Cycle 19: number analyzed (Participants) | 6
  Cycle 19 | 0.3 (0.64)
  Cycle 20: number analyzed (Participants) | 4
  Cycle 20 | 0.2 (0.37)
  Cycle 21: number analyzed (Participants) | 3
  Cycle 21 | 0.0 (0.00)
  Cycle 22: number analyzed (Participants) | 1
  Cycle 22 | 0.0 (NA) — Not applicable = Null value
  Cycle 23: number analyzed (Participants) | 1
  Cycle 23 | 0.0 (NA) — Not applicable = Null value
  Cycle 24: number analyzed (Participants) | 1
  Cycle 24 | 0.0 (NA) — Not applicable = Null value
  Cycle 25: number analyzed (Participants) | 1
  Cycle 25 | 0.0 (NA) — Not applicable = Null value
  Cycle 26: number analyzed (Participants) | 1
  Cycle 26 | 0.0 (NA) — Not applicable = Null value
  Cycle 27: number analyzed (Participants) | 1
  Cycle 27 | 0.0 (NA) — Not applicable = Null value

6. Secondary Outcome: The Number of Units of Red Blood Cell (RBC) Transfusions by Cycle
Description: The number of units of RBC received 56 days prior to treatment, considered the baseline period (baseline period defined as the screening period before the date of the first dose of azacitidine; any laboratory and blood transfusion data reported on the day of the first dose of azacitidine was considered to be baseline data) and during study was standardized per 28 days and summarized by cycle for RBC. The formula for standardizing per 28 days was: [(# of transfusions in the measurement period / length of the measurement period (days)) x 28], where the measurement period was either baseline or the relevant cycle length.
Time Frame: as for outcome 4
Population: ITT includes all participants who were enrolled into the study
Measure: Mean (Standard Deviation); unit: Units of RBC Transfusions
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
Units of RBC Transfusions
  Baseline N = 72 | 2.3 (3.55)
  Overall Post-Baseline Average N = 72 | 3.5 (3.88)
  Overall Change from Baseline N = 72 | 1.2 (4.34)
  Cycle 1 N = 72 | 3.6 (3.41)
  Cycle 2: number analyzed (Participants) | 66
  Cycle 2 | 3.6 (4.88)
  Cycle 3: number analyzed (Participants) | 59
  Cycle 3 | 3.0 (3.68)
  Cycle 4: number analyzed (Participants) | 56
  Cycle 4 | 2.7 (3.73)
  Cycle 5: number analyzed (Participants) | 50
  Cycle 5 | 2.5 (3.94)
  Cycle 6: number analyzed (Participants) | 46
  Cycle 6 | 2.0 (3.46)
  Cycle 7: number analyzed (Participants) | 39
  Cycle 7 | 1.7 (3.84)
  Cycle 8: number analyzed (Participants) | 36
  Cycle 8 | 1.7 (2.68)
  Cycle 9: number analyzed (Participants) | 31
  Cycle 9 | 0.9 (1.56)
  Cycle 10: number analyzed (Participants) | 29
  Cycle 10 | 1.2 (2.25)
  Cycle 11: number analyzed (Participants) | 28
  Cycle 11 | 1.3 (1.97)
  Cycle 12: number analyzed (Participants) | 24
  Cycle 12 | 1.1 (2.21)
  Cycle 13: number analyzed (Participants) | 17
  Cycle 13 | 1.2 (2.62)
  Cycle 14: number analyzed (Participants) | 15
  Cycle 14 | 0.4 (1.05)
  Cycle 15: number analyzed (Participants) | 13
  Cycle 15 | 1.1 (2.07)
  Cycle 16: number analyzed (Participants) | 10
  Cycle 16 | 0.9 (1.61)
  Cycle 17: number analyzed (Participants) | 7
  Cycle 17 | 1.2 (3.28)
  Cycle 18: number analyzed (Participants) | 7
  Cycle 18 | 1.6 (3.07)
  Cycle 19: number analyzed (Participants) | 6
  Cycle 19 | 0.8 (1.37)
  Cycle 20: number analyzed (Participants) | 4
  Cycle 20 | 1.1 (1.42)
  Cycle 21: number analyzed (Participants) | 3
  Cycle 21 | 0.4 (0.62)
  Cycle 22 N: number analyzed (Participants) | 1
  Cycle 22 N | 0 (NA) — Not applicable= Null value
  Cycle 23: number analyzed (Participants) | 1
  Cycle 23 | 0.0 (NA) — Not applicable= Null value
  Cycle 24: number analyzed (Participants) | 1
  Cycle 24 | 0.0 (NA) — Not applicable= Null value
  Cycle 25: number analyzed (Participants) | 1
  Cycle 25 | 0.0 (NA) — Not applicable= Null value
  Cycle 26: number analyzed (Participants) | 1
  Cycle 26 | 0.0 (NA) — Not applicable= Null value
  Cycle 27: number analyzed (Participants) | 1
  Cycle 27 | 0.0 (NA) — Not applicable= Null value

7. Secondary Outcome: The Number of RBC Transfusions by Cycle
Description: The number of RBC transfusions received 56 days prior to treatment, considered the baseline period (baseline period defined as the screening period before the date of the first dose of azacitidine; any laboratory and blood transfusion data reported on the day of the first dose of azacitidine was considered to be baseline data) and during study was standardized per 28 days and summarized by cycle for platelets. The formula for standardizing per 28 days was: [(# of transfusions in the measurement period / length of the measurement period (days)) x 28], where the measurement period was either baseline or the relevant cycle length.
Time Frame: as for outcome 4
Population: Intent to Treat (ITT) includes all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: RBC Transfusions
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
RBC Transfusions
  Baseline N = 72 | 1.1 (1.79)
  Overall Post-Baseline Average N = 72 | 1.6 (1.97)
  Overall Change from Baseline N = 72 | 0.5 (2.12)
  Cycle 1 N = 72 | 1.7 (1.64)
  Cycle 2: number analyzed (Participants) | 66
  Cycle 2 | 1.7 (2.56)
  Cycle 3: number analyzed (Participants) | 59
  Cycle 3 | 1.4 (1.81)
  Cycle 4: number analyzed (Participants) | 56
  Cycle 4 | 1.2 (1.73)
  Cycle 5: number analyzed (Participants) | 50
  Cycle 5 | 1.1 (1.81)
  Cycle 6: number analyzed (Participants) | 46
  Cycle 6 | 0.9 (1.63)
  Cycle 7: number analyzed (Participants) | 39
  Cycle 7 | 0.8 (1.97)
  Cycle 8: number analyzed (Participants) | 36
  Cycle 8 | 0.8 (1.23)
  Cycle 9: number analyzed (Participants) | 31
  Cycle 9 | 0.4 (0.74)
  Cycle 10: number analyzed (Participants) | 29
  Cycle 10 | 0.5 (0.94)
  Cycle 11: number analyzed (Participants) | 28
  Cycle 11 | 0.5 (0.78)
  Cycle 12: number analyzed (Participants) | 24
  Cycle 12 | 0.4 (0.87)
  Cycle 13: number analyzed (Participants) | 17
  Cycle 13 | 0.5 (0.94)
  Cycle 14: number analyzed (Participants) | 15
  Cycle 14 | 0.2 (0.53)
  Cycle 15: number analyzed (Participants) | 13
  Cycle 15 | 0.4 (0.77)
  Cycle 16: number analyzed (Participants) | 10
  Cycle 16 | 0.4 (0.57)
  Cycle 17: number analyzed (Participants) | 7
  Cycle 17 | 0.3 (0.91)
  Cycle 18: number analyzed (Participants) | 7
  Cycle 18 | 0.7 (1.17)
  Cycle 19: number analyzed (Participants) | 6
  Cycle 19 | 0.4 (0.64)
  Cycle 20: number analyzed (Participants) | 4
  Cycle 20 | 0.6 (0.71)
  Cycle 21: number analyzed (Participants) | 3
  Cycle 21 | 0.2 (0.31)
  Cycle 22: number analyzed (Participants) | 1
  Cycle 22 | 0.0 (NA) — Not applicable= Null value
  Cycle 23: number analyzed (Participants) | 1
  Cycle 23 | 0.0 (NA) — Not applicable= Null value
  Cycle 24: number analyzed (Participants) | 1
  Cycle 24 | 0.0 (NA) — Not applicable= Null value
  Cycle 25: number analyzed (Participants) | 1
  Cycle 25 | 0.0 (NA) — Not applicable= Null value
  Cycle 26: number analyzed (Participants) | 1
  Cycle 26 | 0.0 (NA) — Not applicable= Null value
  Cycle 27: number analyzed (Participants) | 1
  Cycle 27 | 0.0 (NA) — Not applicable= Null value

8. Secondary Outcome: The Number of Infections (Post-baseline Average) Requiring Intravenous (IV) Antibiotics, Anti-fungals, or Antivirals by Cycle
Description: The on-treatment adverse event of infection requiring IV antibiotics, antifungals, or antivirals per 28 days/cycle. The overall post-baseline average is the average of number of infections requiring IV antibiotics or IV antiviral per 28 days/cycle.
Time Frame: as for outcome 4
Population: Intent to Treat (ITT) includes all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: Infections
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
Infections
  Baseline N = 72 | 0.0 (0.20)
  Overall Post Baseline Average N = 72 | 0.6 (1.43)
  Overall Change from Baseline N =72 | 0.5 (1.45)
  Cycle 1 N = 72 | 0.6 (1.32)
  Cycle 2: number analyzed (Participants) | 66
  Cycle 2 | 0.5 (1.67)
  Cycle 3: number analyzed (Participants) | 59
  Cycle 3 | 0.4 (0.86)
  Cycle 4: number analyzed (Participants) | 56
  Cycle 4 | 0.5 (1.03)
  Cycle 5: number analyzed (Participants) | 50
  Cycle 5 | 0.4 (0.72)
  Cycle 6: number analyzed (Participants) | 46
  Cycle 6 | 0.2 (0.61)
  Cycle 7: number analyzed (Participants) | 39
  Cycle 7 | 0.3 (1.01)
  Cycle 8: number analyzed (Participants) | 36
  Cycle 8 | 0.2 (0.47)
  Cycle 9: number analyzed (Participants) | 31
  Cycle 9 | 0.1 (0.32)
  Cycle 10: number analyzed (Participants) | 29
  Cycle 10 | 0.2 (0.44)
  Cycle 11: number analyzed (Participants) | 28
  Cycle 11 | 0.1 (0.31)
  Cycle12: number analyzed (Participants) | 24
  Cycle12 | 0.1 (0.27)
  Cycle 13: number analyzed (Participants) | 17
  Cycle 13 | 0.1 (0.24)
  Cycle 14 15: number analyzed (Participants) | 15
  Cycle 14 15 | 0.1 (0.32)
  Cycle 15: number analyzed (Participants) | 13
  Cycle 15 | 0.3 (0.70)
  Cycle 16: number analyzed (Participants) | 10
  Cycle 16 | 0.3 (0.42)
  Cycle 17: number analyzed (Participants) | 7
  Cycle 17 | 0.4 (0.75)
  Cycle 18: number analyzed (Participants) | 7
  Cycle 18 | 0.4 (0.74)
  Cycle 19: number analyzed (Participants) | 6
  Cycle 19 | 0.2 (0.41)
  Cycle 20: number analyzed (Participants) | 4
  Cycle 20 | 0.0 (0.00)
  Cycle 21: number analyzed (Participants) | 3
  Cycle 21 | 0.0 (0.00)
  Cycle 22: number analyzed (Participants) | 1
  Cycle 22 | 0.9 (NA) — Not Applicable = Null value
  Cycle 23: number analyzed (Participants) | 1
  Cycle 23 | 1.0 (NA) — Not Applicable = Null value
  Cycle 24: number analyzed (Participants) | 1
  Cycle 24 | 0.0 (NA) — Not Applicable = Null value
  Cycle 25: number analyzed (Participants) | 1
  Cycle 25 | 0.0 (NA) — Not Applicable = Null value
  Cycle 26 N: number analyzed (Participants) | 1
  Cycle 26 N | 0.0 (NA) — Not Applicable = Null value
  Cycle 27: number analyzed (Participants) | 1
  Cycle 27 | 0.0 (NA) — Not Applicable = Null value

9. Secondary Outcome: Kaplan Meier Estimates for Overall Survival (OS)
Description: Overall survival is defined as time to death from any cause, is calculated using date of first dose and date of death, or date of last follow-up for censored participants. Those, who die regardless of the cause of death, will be considered to have an event.
Time Frame: Until the end of the survival follow-up period; Up to data cut-off of 29 January 2015; 894 days
Population: Intent to Treat (ITT) includes all participants who were enrolled into the study.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
months
  Median OS | 22.0 [15.1 to NA] — The data for overall survival has not matured and does not exist as of data cut- off date of 29 Jan 2015 as the study is on-going
  25th percentile OS | 8.5 [6.1 to 13.8]
  75th Percentile OS | NA [24.2 to NA] — The data for overall survival among the 75th percentile has not matured and does not exist as of data cut-off date of 29 Jan 2015 as the study is on-going. This also applies to the upper limit.

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During the Parent Phase
Description: A treatment-emergent adverse events (TEAE) was defined as AEs with an onset date on or after the date of first dose and within 28 days after the date of the last dose. Any AE that occurred beyond this timeframe and was assessed by the investigator as possibly related to study drug was considered treatment-emergent. The intensity and severity of AEs was assessed by the investigator according to the Common Terminology Criteria for Adverse Event (CTCAE) Version 4.0. For any AEs not listed in the CTCAE grading system, the intensities of these events was assessed by the Investigator using the 5-point scale: Grade 1 = Mild, Grade 2 = Moderate; Grade 3 = Severe, Grade 4 = Life threatening, Grade 5 = Death. An SAE is any AE occurring that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, and constitutes an important medical event.
Time Frame: Up to 29 January 2015; from the first dose of study drug to 28 days after the date of the last dose of study drug (maximum time on study was 244 days)
Population: Safety population included all participants who received at least one dose of azacitidine and had at least one post-dose safety assessment
Measure: Number; unit: participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 72
participants
  ≥ 1 TEAE | 72
  ≥ 1 Grade 3 or 4 TEAE | 70
  ≥ 1 TEAE related to study drug | 68
  ≥ 1 Grade 3 or 4 TEAE related to study drug | 59
  ≥ 1 serious TEAE | 38
  ≥ 1 Grade 3 or 4 serious TEAE | 33
  ≥ 1 serious TEAE related to study drug | 28
  ≥ 1 TEAE leading to discontinuation of study drug | 14
  ≥ 1 TEAE leading to dose reduction of study drug | 19
  ≥1 TEAE leading to dose interruption of study drug | 49
  ≥1 TEAE leading to dose reduction/interruption | 50
  ≥1 TEAE with outcome of death | 11

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC∞) of Azacitidine
Description: Area under the plasma concentration-time curve from time zero to infinity (AUC∞) following multiple doses of Azacitidine on Day 7; if possible, the area under the concentration-time curve from time zero to infinity, calculated by the linear trapezoidal rule and extrapolated to infinity was calculated according to the following equation: AUC∞ = AUCt + (Ct/ λz ), where Ct is the last quantifiable concentration. No AUC extrapolation will be performed with unreliable λz. If % AUC extrapolated is ≥ 25%, AUC∞ will not be reported
Time Frame: PK blood samples collected at 0.25, 0.5, 1,2,3,4, 6 and 8 hours after azacitidine administration on Day 7
Population: The PK population includes up to 12 participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
ng*h/mL | 1172.6 (18.0)

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUCt) of Azacitidine
Description: Area under the plasma concentration-time curve from time zero to the last quantifiable time point, calculated by the linear trapezoidal rule when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing.
Time Frame: PK blood samples collected at 0.25, 0.5, 1,2,3,4, 6 and 8 hours after azacitidine administration on Day 7
Population: The PK population includes up to 12 participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
ng*h/mL | 1161.9 (17.7)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Azacitidine
Description: The observed maximum plasma concentration obtained directly from the observed concentration versus time data.
Time Frame: PK blood samples collected at 0.25, 0.5, 1,2,3,4, 6 and 8 hours after azacitidine administration on Day 7
Population: The PK population includes up to 12 participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
ng/mL | 1264.6 (30.7)

14. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Azacitidine
Description: Time to maximum observed plasma concentration obtained directly from the observed concentration versus time data.
Time Frame: PK blood samples collected at 0.25, 0.5, 1,2,3,4, 6 and 8 hours after azacitidine administration on Day 7
Population: The PK population includes up to 12 participants with evaluable azacitidine plasma PK profile.
Measure: Median (Full Range); unit: hours
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
hours | 0.25 (27.66) [0.23 to 0.50]

15. Secondary Outcome: Terminal Phase of Half-life (T1/2) of Azacitidine
Description: The apparent terminal half-life was calculated according to the following equation t½ = 0.693/λz.
Time Frame: PK blood samples collected at 0.25, 0.5, 1,2,3,4, 6 and 8 hours after azacitidine administration on Day 7
Population: The PK population includes up to 12 participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
hours | 0.8 (69.0)

16. Secondary Outcome: Apparent Total Plasma Clearance (CL/F) of Azacitidine
Description: Apparent total plasma clearance (CL/F) of Azacitidine was calculated as Dose/AUC∞
Time Frame: PK blood samples collected at 0.25, 0.5, 1,2,3,4, 6 and 8 hours after azacitidine administration on Day 7
Population: The PK population includes up to 12 participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hours
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
Liters/hours | 107.2 (19.1)

17. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of Azacitidine
Description: Apparent volume of distribution, was calculated according to the equation: Vd/F = (CL/F)/λz
Time Frame: PK blood samples collected at 0.25, 0.5, 1,2,3,4, 6 and 8 hours after azacitidine administration on Day 7
Population: The PK population includes up to 12 participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
Liters | 121.5 (65.1)

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During the Extension Phase
Description: as for outcome 10
Time Frame: Up to final data cut off date of 25 April 2018; from the first dose of study drug extesnion of 29 December 2014 to 28 days after the date of the last dose of study drug; median duration of any dose of study drug was 169 days
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 15
participants
  ≥ 1 TEAE | 14
  ≥ 1 TEAE related to study drug | 8
  ≥ 1 Grade 3 or 4 TEAE | 13
  ≥ 1 Grade 3 or 4 TEAE related to study drug | 6
  ≥ 1 serious TEAE | 5
  ≥ 1 serious TEAE related to study drug | 1
  ≥ 1 Grade 3 or 4 serious TEAE | 5
  ≥1 TEAE leading to dose interruption of study drug | 4
  ≥1 TEAE leading to dose reduction/interruption | 4

ADVERSE EVENTS:
Time Frame: Azacitidine Exposure across all cycles: median duration of azacitidine treatment was 786 days (range 428 to 1507).
Description: For extension phase: From 29 December 2014 to 28 days after the date of the last dose of study drug; median treatment duration of any dose of azacitidine was 169 days; range: 7 to 1112 days.
Groups:
- Azacitidine - Parent Phase: Azacitidine 75 mg/m^2/day subcutaneously (SC) for 7 days every 28 days until disease progression (DP), adverse events (AE), withdrawal of consent from further treatment, withdrawal of consent, death, lost to follow-up, or protocol violation.
- Azacitdine - Extension Phase: Azacitidine 75 mg/m^2/day subcutaneously for 7 days every 28 days until disease progression (DP), adverse events (AE), withdrawal of consent from further treatment, withdrawal of consent, death, lost to follow-up, or protocol violation
Arm/Group | Azacitidine - Parent Phase | Azacitdine - Extension Phase
All-Cause Mortality (participants affected / at risk) | 13/72 | 0/15
Serious Adverse Events (participants affected / at risk) | 38/72 | 5/15
Other Adverse Events (participants affected / at risk) | 72/72 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine - Parent Phase (N=72) | Azacitdine - Extension Phase (N=15)
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 4 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Anal abscess (Infections and infestations) | 1 | 0
Anal infection (Infections and infestations) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Cellulitis (Infections and infestations) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Fungal sepsis (Infections and infestations) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gingival infection (Infections and infestations) | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lung infection (Infections and infestations) | 2 | 2
Mouth haemorrhage (Gastrointestinal disorders) | 3 | 0
Myelitis (Infections and infestations) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonia (Infections and infestations) | 11 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 3 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0
Erythropenia (Blood and lymphatic system disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal Failure, Acute (Renal and urinary disorders) | 0 | 1
Henoch-Schonlein Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine - Parent Phase (N=72) | Azacitdine - Extension Phase (N=15)
Abdominal discomfort (Gastrointestinal disorders) | 8 | 2
Abdominal distension (Gastrointestinal disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Alanine aminotransferase increased (Investigations) | 10 | 2
Anaemia (Blood and lymphatic system disorders) | 38 | 6
Aspartate aminotransferase increased (Investigations) | 6 | 2
Asthenia (General disorders) | 6 | 3
Cellulitis (Infections and infestations) | 4 | 0
Conjunctival haemorrhage (Eye disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 22 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 15 | 3
Dizziness (Nervous system disorders) | 5 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Fatigue (General disorders) | 4 | 0
Gingival bleeding (Gastrointestinal disorders) | 8 | 1
Gingival infection (Infections and infestations) | 5 | 0
Gingivitis (Infections and infestations) | 16 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 12 | 0
Leukopenia (Blood and lymphatic system disorders) | 48 | 10
Lung infection (Infections and infestations) | 8 | 1
Mouth ulceration (Gastrointestinal disorders) | 6 | 0
Nausea (Gastrointestinal disorders) | 19 | 3
Neutropenia (Blood and lymphatic system disorders) | 48 | 6
Oedema peripheral (General disorders) | 9 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Pneumonia (Infections and infestations) | 19 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Purpura (Skin and subcutaneous tissue disorders) | 5 | 0
Pyrexia (General disorders) | 21 | 2
Skin infection (Infections and infestations) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 52 | 10
Toothache (Gastrointestinal disorders) | 4 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 27 | 1
Vomiting (Gastrointestinal disorders) | 15 | 0
Weight decreased (Investigations) | 12 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Localized Oedema (General disorders) | 0 | 1
Nodule (General disorders) | 0 | 1
Hepatic Stenosis (Hepatobiliary disorders) | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Soft Tissue Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Bilirubin Conjugated Increased (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 1
Blood Fibrinogen Decreased (Investigations) | 0 | 1
Blood Urea Increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemoglobinuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally sixty (60) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.